CLINICAL TRIAL: NCT06891521
Title: Electroacupuncture for Preventing Adverse Events Associated With Cancer Immunotherapy: A Prospective, Multicenter, Open-Label, Single-Arm Clinical Study
Brief Title: Electroacupuncture for Preventing Adverse Events of Cancer Immunotherapy
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Qinghai Red Cross Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: QRCH-2025002
Record Dates: First submitted 2025-02-27; First posted 2025-03-24 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Cancer; Adverse Events
Keywords: Electroacupuncture; immunotherapy; immune-related adverse events (irAEs); malignant tumors
MeSH Terms: conditions — Neoplasms | interventions — Electroacupuncture

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Electroacupuncture group (Experimental): Patients received electroacupuncture therapy on the day before and the first day of each ICIs treatment cycle. Intervention: The patient received electroacupuncture and standard antitumor therapy.
  Interventions: Procedure: Electroacupuncture

INTERVENTIONS:
Procedure: Electroacupuncture — Patients received electroacupuncture on the day before and the first day of each ICIs treatment cycle. The electroacupuncture points selected Zusanli (ST36), Quchi (LI11), and Hegu (LI4). Patients will be positioned supine, and the acupuncturist will disinfect the local skin at the acupuncture points using 75% ethanol on cotton balls. A disposable acupuncture needle (0.3mm × 40mm) will be inserted using either a single-hand or double-hand needling technique, with rapid, direct insertion. Once the needle reaches a depth of approximately 0.5 cun, the technique of lifting, thrusting, twirling, and rotating will be applied. After obtaining "de qi", the needles will be retained for 30 minutes. Needling will be performed once every 10 minutes, and the needling technique used will be a balanced reinforcing and reducing method. Electroacupuncture will be applied using a dense-wave form, with a frequency of 2 Hz and an intensity not exceeding 10 mA.

SUMMARY:
This study aims to investigate the preventive effects of electroacupuncture on immune-related adverse events (irAEs) in patients with malignant solid tumors at the neoadjuvant stage, locally advanced, unresectable, or metastatic stages, who are receiving immune checkpoint inhibitors (ICIs) monotherapy, ICIs combined with anti-angiogenic agents, or ICIs combined with chemotherapy. The study will evaluate the efficacy, safety and mechanisms of electroacupuncture in preventing irAEs in a multicenter setting.

DETAILED DESCRIPTION:
This study is a prospective, multicenter, open-label, single-arm clinical trial aimed at collecting data from patients with malignant solid tumors at the neoadjuvant stage, locally advanced, unresectable, or metastatic stages, who are receiving immune checkpoint inhibitors (ICIs) monotherapy, ICIs combined with anti-angiogenic agents, or ICIs combined with chemotherapy. The objective is to evaluate the efficacy and safety of electroacupuncture in preventing immune-related adverse events (irAEs). Patients who meet the inclusion and exclusion criteria will be formally enrolled after screening and providing informed consent. Eligible patients will receive electroacupuncture treatment, with the intervention occurring on the day before and the first day of each ICIs treatment cycle. During the treatment period, the incidence, severity, and timing of irAEs will be monitored through follow-up assessments. Additionally, questionnaires will be collected to evaluate the impact of electroacupuncture on quality of life. Blood samples will be collected for analysis of changes in inflammatory cytokines and peripheral blood lymphocyte subset proportions. The study will also assess primary and secondary outcomes, as well as adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years, any gender, any nationality.
2. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
3. A definitive diagnosis of malignant tumor confirmed by pathology, and no previous treatment with PD-1/PD-L1 inhibitors.
4. Patients who are receiving their first treatment with PD-1/PD-L1 inhibitors monotherapy, PD-1/PD-L1 inhibitors combined with anti-angiogenic agents, or combined chemotherapy.
5. Expected survival of more than 3 months.
6. Normal bone marrow and organ function.
7. Premenopausal women must use adequate contraception.
8. Written informed consent obtained from the patient prior to enrollment.

Exclusion Criteria:

1. Patients who have previously received or are currently receiving immunotherapy monotherapy, immunotherapy combined with chemotherapy, or immunotherapy combined with targeted therapy.
2. Patients who have undergone acupuncture, radiotherapy, or surgery within 4 weeks prior to the start of treatment.
3. Patients who have received any dose of systemic corticosteroid treatment within 72 hours prior to Day 1 of Cycle 1.
4. Patients with active systemic autoimmune diseases within the past 2 years (such as but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hepatitis, pituitaryitis, vasculitis, nephritis, hyperthyroidism, hypothyroidism; subjects with a history of vitiligo or asthma in childhood who have been in complete remission with no intervention in adulthood may be included; subjects requiring bronchodilator medical intervention should be excluded), diagnosed with immunodeficiency or treated with immunosuppressive therapy within the past week, human immunodeficiency virus (HIV) (+), history of non-infectious pneumonia treated with glucocorticoids, pneumonia, active tuberculosis, active hepatitis B or C virus infection, or currently undergoing any systemic treatment for active infections.
5. Significant abnormal laboratory values (platelet count, absolute neutrophil count, free triiodothyronine (FT3), free thyroxine (FT4), thyroid stimulating hormone(TSH), adrenocorticotropic hormone (ACTH), morning cortisol, glycated hemoglobin (HbA1c), C-peptide, autoantibodies, alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase, prothrombin time/international normalized ratio (PT/INR), serum bilirubin, amylase, lipase, CRP).
6. Skin diseases or inflammatory skin reactions that may interfere with clinical trial outcomes.
7. Patients who have developed lymphedema at the site of acupuncture stimulation after receiving any acupuncture treatment.
8. Patients who fear electroacupuncture stimulation or are allergic to stainless steel needles.
9. Patients with psychiatric disorders, or those taking any antipsychotic or antidepressant medications.
10. Any unresolved skin toxicity caused by previous chemotherapy or radiotherapy, except for hair loss.
11. Patients with diabetes.
12. Any other diseases, metabolic disorders, physical examination results, or clinical laboratory findings that raise reasonable suspicion of a disease or condition that may affect the interpretation of the outcomes or put the participant at high risk for treatment complications.
13. Pregnant or breastfeeding women, or women planning to become pregnant during the study period.
14. Severe medical or psychiatric conditions.
15. Any patient deemed unsuitable for enrollment by the investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Estimated)
Dates: Start 2025-03-20 (Estimated); Primary Completion 2027-03-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
The overall incidence of any grade of immune-related adverse events (irAEs). | 48 weeks.
  IrAEs are defined as any adverse events potentially related to immune mechanisms that occur during or after ICIs treatment. Adverse events will be assessed using the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.

SECONDARY OUTCOMES:
The incidence of Grade ≥3 immune-related adverse events (irAEs). | 48 weeks.
  IrAEs are defined as any adverse events potentially related to immune mechanisms that occur during or after ICIs treatment. Adverse events will be assessed using the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
The time to onset of Grade ≥3 immune-related adverse events (irAEs). | 48 weeks.
  The time to onset is defined as the period from the initiation of immune checkpoint inhibitor (ICIs) treatment to the occurrence of the immune-related adverse event. Adverse events will be assessed using the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
The time to onset of any grade of immune-related adverse events (irAEs). | 48 weeks.
  The time to onset is defined as the period from the initiation of immune checkpoint inhibitor (ICIs) treatment to the occurrence of the immune-related adverse event. Adverse events will be assessed using the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
The incidence of any grade and Grade ≥3 immune-related adverse events (irAEs) associated with ICIs combination therapy. | 48 weeks.
  IrAEs are defined as any adverse events potentially related to immune mechanisms that occur during or after ICIs treatment. Adverse events will be assessed using the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
The incidence of any grade and Grade ≥3 treatment-related adverse events (TRAEs) associated with ICIs combined with chemotherapy. | 48 weeks.
  TRAEs are defined as any adverse events caused by ICIs combined with chemotherapy during or after the treatment period. Adverse events will be assessed using the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
The incidence of any grade and Grade ≥3 immune-related adverse events (irAEs) associated with ICIs monotherapy. | 48 weeks.
  IrAEs are defined as any adverse events potentially related to immune mechanisms that occur during or after ICIs treatment. Adverse events will be assessed using the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
The incidence of any grade and Grade ≥3 treatment-related adverse events (TRAEs) associated with ICIs combined with anti-angiogenic agents. | 48 weeks.
  TRAEs are defined as any adverse events caused by ICIs combined with anti-angiogenic agents during or after the treatment period. Adverse events will be assessed using the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
The incidence of any grade and Grade ≥3 hyperthyroidism and hypothyroidism. | 48 weeks.
  Adverse events will be assessed using the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
The incidence of any grade and Grade ≥3 rash. | 48 weeks.
  Adverse events will be assessed using the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
The incidence of any grade and Grade ≥3 hepatitis. | 48 weeks.
  Adverse events will be assessed using the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
The incidence of any grade and Grade ≥3 pneumonia. | 48 weeks.
  Adverse events will be assessed using the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
The incidence of any grade and Grade ≥3 abnormal blood glucose levels. | 48 weeks.
  Adverse events will be assessed using the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Comparison of biomarker changes before and after electroacupuncture treatment. | 48 weeks.
  The differences in biomarkers will be monitored through hematological parameters, including: inflammatory biomarkers such as C-reactive protein (CRP), procalcitonin (PCT), inflammatory cytokines like IL-1β, IL-6, IL-10, TNF-α, IFN-γ, and changes in the proportions of peripheral blood lymphocyte subsets (CD4+, CD8+ T cells, natural killer cells (NK cells), regulatory T cells (Treg cells), and myeloid-derived suppressor cells (MDSCs)), as well as tumor markers.
The incidence of adverse events related to electroacupuncture treatment. | 48 weeks.
  Adverse events will be assessed using the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 to determine the proportion of side effects associated with electroacupuncture.
The evaluation of the difference in quality of life before and after electroacupuncture treatment. | 48 weeks.
  Quality of life will be assessed using the EuroQol Five-Dimensional Questionnaire (EQ-5D-5L). EQ-5D-5L is a standardized tool for assessing health-related quality of life, which includes five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has five levels describing an individual's functional or well-being status in a specific area. Additionally, the EQ-5D-5L includes a visual analogue scale, allowing individuals to rate their overall health status on a scale from 0 (worst health) to 100 (best health).
16.Adherence to electroacupuncture treatment. | 48 weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- Qinghai, China, Qinghai Red Cross Hospital, Xining, Qinghai, China